CLINICAL TRIAL: NCT00995202
Title: Follow-Up of Fully Resected Stage II or III Colorectal Cancer. Phase III Multicentric Prospective Randomised Study
Brief Title: Follow-Up Care With or Without CEA Assessments in Patients Who Have Undergone Surgery for Stage II or Stage III Colorectal Cancer
Acronym: SURVEILLANCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: PRODIGE 13; FFCD-PRODIGE-13; 2009-A00536-51; EU-20979
Record Dates: First submitted 2009-10-14; First posted 2009-10-15 (Estimated); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Colorectal Cancer
Keywords: stage II colon cancer; stage II rectal cancer; stage III colon cancer; stage III rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: This study is a surveillance study not an interventional study with products
Oversight: Data Monitoring Committee: No

ARMS (4):
- Standard Monitoring CEA/ Standard Imagery (Other): No specific follow-up of CEA and Standard imagery
  Interventions: Procedure: Standard Monitoring CEA; Procedure: Standard Monitoring Imagery
- Intensive monitoring CEA/ Standard Imagery (Other): Intensive follow-up CEA and Standard imagery .
  Interventions: Procedure: Intensive Monitoring CEA; Procedure: Standard Monitoring Imagery
- Intensive Monitoring CEA / Intensive Monitoring Imagery (Other): Intensive follow-up CEA and Intensive imagery
  Interventions: Procedure: Intensive Monitoring CEA; Procedure: Intensive Monitoring Imagery
- Standard Monitoring CEA/ Intensive Monitoring Imagery (Other): No specific follow-up of CEA and Intensive Imagery
  Interventions: Procedure: Standard Monitoring CEA; Procedure: Intensive Monitoring Imagery

INTERVENTIONS:
Procedure: Standard Monitoring CEA — No specific follow-up of CEA
  Arms: Standard Monitoring CEA/ Intensive Monitoring Imagery; Standard Monitoring CEA/ Standard Imagery
Procedure: Intensive Monitoring CEA — CEA levels are measured every 3 months for 3 years, then every 6 months for 2 years.
  Arms: Intensive Monitoring CEA / Intensive Monitoring Imagery; Intensive monitoring CEA/ Standard Imagery
Procedure: Standard Monitoring Imagery — Abdominal ultrasound examination every 3 months during 3 years then every 6 months during 2 years then annually. Chest X-ray examination eveyr 6 months during 3 years then annually during 2 years
  Arms: Intensive monitoring CEA/ Standard Imagery; Standard Monitoring CEA/ Standard Imagery
Procedure: Intensive Monitoring Imagery — Alternation every 3 months of TDM thoraco-abdomino-pelvis and abdominal ultrasound examination during 3 years and twice a year after during 2 years. Coloscopy at 3 years and then evry 5 years if normal
  Arms: Intensive Monitoring CEA / Intensive Monitoring Imagery; Standard Monitoring CEA/ Intensive Monitoring Imagery

SUMMARY:
RATIONALE: Diagnostic procedures, such as ultrasound, x-ray, colonoscopy, CT scan, and CEA assessment, may help monitor a patient's response to surgery. It is not yet known which follow-up regimen is more effective in patients who have undergone surgery for colorectal cancer.

PURPOSE: This randomized phase III trial is comparing two types of follow-up care with or without CEA assessments to see how well they work in patients who have undergone surgery for stage II or stage III colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the efficacy of reinforced versus standard follow-up care and the utility of follow-up CEA assessments in patients with fully resected stage II or III colorectal cancer.

OUTLINE: This is a multinational/multicenter study. Patients are randomized to 1 of 2 follow-up arms.

* Standard follow-up: Patients undergo clinical assessments every 3 months until year 3 and every 6 months until year 5. They are then assessed at least yearly thereafter. Patients undergo abdominal ultrasound every 3 months until year 3 and then every 6 months until year 5; chest x-ray every 6 months until year 3 and then annually until year 5; and colonoscopy at 3 years after surgery then every 3 to 6 years thereafter.
* Reinforced follow-up: Patients undergo clinical assessments every 3 months until year 3 and every 6 months until year 5. They are then assessed at least yearly thereafter. Patients undergo alternate assessments every 3 months comprising thoraco-abdomino-pelvic CT scan or abdominal ultrasound until year 3 and then every 6 months until year 5. They also undergo colonoscopy at 3 years after surgery then every 3 to 6 years thereafter.

Patients undergo a second randomization to 1 of 2 follow-up arms at the beginning of the study.

* CEA measurement: Patients undergo measurement of CEA levels every 3 months until year 3, every 6 months until year 5, and at least yearly thereafter.
* No CEA measurement: Patients do not undergo CEA measurement. Blood and tissue blocks of normal and tumor tissues are collected for the validation of protein serum, genetics, or immunologic markers predictive for relapse.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologically confirmed adenocarcinoma of the colon or rectum

  * Stage II or III disease
  * No distant metastatic disease
* Has undergone curative resection for no residual tumor
* Carcinoembryonic antigen (CEA) ≤ 1.5 x upper limit of normal after surgery

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No inflammatory bowel disease
* No other malignancy within the past 5 years except basal cell carcinoma of the skin and/or carcinoma in situ of the cervix
* No genetic syndromes

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1997 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Overall survival rate | 5 years
  Time between randomization and date of death (all causes)

SECONDARY OUTCOMES:
Disease-free survival rate | 5 years
  Time between randomization and first recurrence (local or metastatic) or death (all causes)

CONTACTS AND LOCATIONS:
Overall Officials: Come Lepage, Pr, Principal Investigator — Centre Hospitalier Universitaire Dijon
Locations (117):
- Clinique Sud Luxembourg, Arlon, Belgium
- France (115):
  - CH, Abbeville
  - Clinique Isabelle, Abbeville
  - CHU Nord, Amiens
  - CHU, Angers
  - CH, Antibes
  - CH, Aubenas
  - CH, Auch
  - CH, Auxerre
  - Polyclinique Ste Marguerite, Auxerre
  - CH Henri Duffaut, Avignon
  - Clinique Sainte Cahterine, Avignon
  - Centre d'oncologie et de radiothérapie du Pays Basque, Bayonne
  - CH, Beaune
  - CH, Beauvais
  - CHU J Minjoz, Besançon
  - Centre de Radiothérapie et d'oncologie médicale, Béziers
  - CH, Béziers
  - CH, Blois
  - CH, Bobigny
  - Polyclinique Nord Aquitaine, Bordeaux
  - CH Duchenne, Boulogne-sur-Mer
  - CH, Bourg-en-Bresse
  - Hôpital du Morvan, Brest
  - CH, Briey
  - CHIC, Castres
  - CH, Challans
  - Hôpital Sainte Marie, Chalon-sur-Saône
  - CH, Chambéry
  - Clinique du Cléret et Clinique Saint Joseph, Chambéry
  - CH, Châlons-en-Champagne
  - CH, Cholet
  - CHU Estaing, Clermont-Ferrand
  - Hôpital Pästeur, Colmar
  - CH, Compiègne
  - Clinique des 2 Caps, Coquelles
  - Clinique des Cèdres, Cornebarrieu
  - Clinique des Acacias, Cucq
  - CH, Dax
  - Cabinet d'HGE - Cours De Gaulle, Dijon
  - Cabinet Privé Point Médical, Dijon
  - Centre d'Oncologie Médicale du Parc, Dijon
  - CHU le bocage, Dijon
  - CH, Draguignan
  - Clinique Saint Vincent, Épernay
  - Centre médical de Forcilles, Férolles-Attilly
  - CHI Saint Raphael, Fréjus
  - CHI, Gap
  - Institut Hollard, Grenoble
  - CH, Haguenau
  - CHD, La Roche-sur-Yon
  - CH, Lagny-sur-Marne
  - CH Louis Pasteur, Le Coudray
  - CH, Le Havre
  - CH, Le Mans
  - Hôpital Robert Boulin, Libourne
  - Centre Oscar Lambret, Lille
  - CHG, Longjumeau
  - Clinique des 4 pavillons, Lormont
  - CHU Lyon Sud, Lyon
  - CH Saint Joseph, Marseille
  - CHU La Timone, Marseille
  - Hôpital Européen, Marseille
  - Hôpital Nord, Marseille
  - CH, Mâcon
  - Polyclinique du Val de Saône, Mâcon
  - Hôpital Layné, Mont-de-Marsan
  - CH, Montbrison
  - CH, Montceau-les-Mines
  - CH, Montélimar
  - CHI Le Raincy Montfermeil, Montfermeil
  - Centre Azuréen de Cancérologie, Mougins
  - Hopital Americain de Paris, Neuilly-sur-Seine
  - Polyclinique Val de Loire, Nevers
  - Hôpital l'Archet II, Nice
  - CHU Carémeau, Nîmes
  - Clinique Valdegour, Nîmes
  - CHR - Sce D'HGE, Orléans
  - CHR - Sce d'Oncologie, Orléans
  - Hôpital Privé Les Peupliers, Paris
  - Hôpital Saint Louis, Paris
  - CH, Pau
  - Centre Catalan d'Oncologie, Perpignan
  - Hôpital Saint Jean, Perpignan
  - CHU Haut Lévèque, Pessac
  - Polyclinique Francheville, Périgueux
  - Centre Hospitalier Annecy Genevois, Pringy
  - CH, Privas
  - CHU Robert Debré, Reims
  - Institut Jean Godinot, Reims
  - CHU Pontchaillou, Rennes
  - CH, Rodez
  - CH Romans, Romans-sur-Isère
  - CH Yves Lefoll, Saint-Brieuc
  - CHPG, Saint-Chamond
  - CH, Saint-Dié
  - CHU, Saint-Etienne
  - Polyclinique Côte Basque Sud, Saint-Jean-de-Luz
  - Centre Joliot Curie, Saint-Martin-Boulogne
  - Clinique de la Côte d'Opale, Saint-Martin-Boulogne
  - Clinique Mutualiste de l'Estuaire - Cité Sanitaire, Saint-Nazaire
  - Clinique, Sainte-Colombe
  - Centre Médical National MGEN Alfred Leune, Sainte-Feyre
  - CH, Semur-en-Auxois
  - CH, Soissons
  - Hôpital Broussais, St-Malo
  - Centre Paul Strauss, Strasbourg
  - Hôpital Sainte Musse, Toulon
  - CH Gustave Dron, Tourcoing
  - CH Trousseau, Tours
  - CH, Valence
  - CHBA, Vannes
  - CH, Vernon
  - CH, Vesoul
  - CH Privé, Villeneuve-d'Ascq
  - CH, Villeneuve-Saint-Georges
- CHU Clarac, Fort-de-France, Martinique

REFERENCES:
- [Background] Lepage C, Phelip JM, Cany L, Faroux R, Manfredi S, Ain JF, Pezet D, Baconnier M, Deguiral P, Terrebone E, Adenis A, Le Malicot K, Bedenne L, Bouche O. Effect of 5 years of imaging and CEA follow-up to detect recurrence of colorectal cancer: The FFCD PRODIGE 13 randomised phase III trial. Dig Liver Dis. 2015 Jul;47(7):529-31. doi: 10.1016/j.dld.2015.03.021. Epub 2015 Apr 2. No abstract available. PMID 25933809